CLINICAL TRIAL: NCT05349214
Title: A Randomized, Double-blind, Placebo Controlled, 3-arm Multicenter Phase 3 Study to Assess the Efficacy and Safety of Ianalumab in Patients With Active Sjogren's Syndrome (NEPTUNUS-2)
Brief Title: Three-arm Study to Assess Efficacy and Safety of Ianalumab (VAY736) in Patients With Active Sjogren's Syndrome
Acronym: NEPTUNUS-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736A2302; 2024-511068-10-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2022-04-08; First posted 2022-04-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sjogren Syndrome
Keywords: Sjogren's syndrome, B-cell depleting, BAFF-R, VAY736, ianalumab, NEPTUNUS
MeSH Terms: conditions — Sjogren's Syndrome | interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, investigator staff, persons performing the assessments and Novartis Clinical Trial Team will remain blinded to the identity of the treatment from the time of randomization until the final database lock
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): ianalumab exposure level 1
  Interventions: Biological: VAY736
- Arm B (Experimental): ianalumab exposure level 2
  Interventions: Biological: VAY736
- Arm C (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAY736 — ianalumab s.c.
  Arms: Arm A; Arm B
Other: Placebo — placebo s.c.
  Arms: Arm C

SUMMARY:
A randomized, double-blind, placebo controlled, 3-arm multicenter phase 3 study to assess the efficacy and safety of ianalumab in patients with active Sjogren's syndrome (NEPTUNUS-2)

DETAILED DESCRIPTION:
Three-arm study of the clinical efficacy, safety and tolerability of ianalumab (VAY736) in patients with active Sjogren's syndrome. The purpose of this study is to demonstrate the clinical efficacy, safety and tolerability of ianalumab (VAY736) administered subcutaneously (s.c.) monthly or every 3 months compared to placebo in patients with active Sjogren's syndrome.

ELIGIBILITY:
Inclusion criteria

* Signed informed consent must be obtained prior to participation in the study
* Women and men ≥ 18 years of age
* Classification of Sjögren's syndrome according to the ACR/EULAR 2016 criteria
* Time since diagnosis of Sjögren's of ≤ 7.5 years at screening
* Positive anti-Ro/SSA antibody at screening

  * Patients negative for anti-Ro/SSA antibody are eligible, if they have a positive salivary gland biopsy confirmed by central expert review
  * Enrollment of anti-Ro/SSA-negative patients will be limited up to ≤10% of the study population
* Screening ESSDAI score of ≥ 5 within the following 8 domains: constitutional, lymphadenopathy, glandular, articular, cutaneous, renal, hematological and biologic.
* Stimulated whole salivary flow (sSF) rate of ≥ 0.05 mL/min at screening
* Ability to communicate well with the Investigator, understand and agree to comply with the requirements of the study
* Patients taking hydroxychloroquine (≤ 400 mg/day), methotrexate (≤ 25 mg/week) or azathioprine (≤ 150 mg/day) alone or in combination, are allowed to continue their medication, and must have been on a stable dose for at least 30 days prior to randomization.
* Patients taking systemic corticosteroids have to be on a stable dose of ≤ 10 mg/day predniso(lo)ne or equivalent for at least 30 days before randomization.
* Patients taking

  * disease-modifying antirheumatic drugs (DMARDs) other than specifically allowed in inclusion criterion #9 or
  * the following Traditional Chinese Medicines: Total glucoside of peony (TGP) or Tripterium glycosides (TG) must discontinue these medications at least 30 days prior to randomization, except for leflunomide, which has to be discontinued for 8 weeks prior to randomization unless a cholestyramine wash-out has been performed.

Exclusion Criteria:

* Presence of another autoimmune rheumatic disease that is active and constitutes the principal illness
* Use of other investigational drugs within 5 half-lives of enrollment, or within 30 days or until the expected pharmacodynamic effect has returned to baseline, whichever is longer3. Prior treatment with ianalumab
* Prior use of a B-cell depleting therapy other than ianalumab within 36 weeks prior to randomization or as long as B-cell count is less than the lower limit of normal or baseline value prior to receipt of previous B cell-depleting therapy (whichever is lower)
* Prior treatment with any of the following:

  1. Within 24 weeks prior to randomization: iscalimab (anti CD-40 mAb), belimumab , abatacept, anti-tumor necrosis factor alpha biologic agents, immunoglobulins plasmapheresis;
  2. Within 12 weeks prior to randomization: i.v. or oral cyclophosphamide, mycophenolate mofetil, i.v. or oral cyclosporine A or any other immunosuppressants (e.g., JAK inhibitors or other kinase inhibitors) unless explicitly allowed by protocol
* Use of corticosteroids (predniso(lo)ne or equivalent corticosteroid) at dose >10 mg/day
* Any one of the following laboratory values at screening:

  * Hemoglobin levels < 8.0 g/dL
  * White blood cells (WBC) count < 2.0 x 10E3/µL
  * Platelet count < 80 x 10E3/µL
  * Absolute neutrophil count (ANC) < 0.8 x 10E3/µL
* Active viral, bacterial or other infections requiring systemic treatment at the time of screening or randomization, or history of recurrent clinically significant infection or of recurrent bacterial infections with encapsulated organisms
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes (e.g., mAb of IgG1 class) or to any of the constituents of the study drug formulation (sucrose, L-histidine hydrochloride/ L-histidine, polysorbate 20)
* History of major organ, hematopoietic stem cell or bone marrow transplant
* Required regular use of medications known to cause dry mouth/eyes as a regular and major side effect, and which have not been on a stable dose for at least 30 days prior to Screening, or any anticipated change in the treatment regimen during the course of the study.
* Use of topical ocular prescription medications (excluding artificial tears, gels, lubricants) that have not been on a stable dose for at least 90 days prior to randomization, or any anticipated change in the treatment regimen during the course of the study
* Receipt of live/attenuated vaccine within a 4-week period prior to randomization
* History of primary or secondary immunodeficiency, including a positive human immunodeficiency virus (HIV) test result
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer or Sjögren's related lymphoma), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* History of sarcoidosis
* Any surgical, medical (e.g., uncontrolled hypertension, heart failure or diabetes mellitus), psychiatric or additional physical condition that the Investigator feels may jeopardize the patient in case of participation in this study
* Chronic infection with hepatitis B (HBV) or hepatitis C (HCV) virus. Positive serology for hepatitis B surface antigen (HBsAg) excludes the subject.

  * HBsAg negative subjects who are hepatitis B core antibody (HBcAb) positive are also excluded unless all of the following criteria are met:

    1. HBV DNA is negative
    2. hepatitis B monitoring is implemented - in these subjects, monthly testing of HBsAg and HBV DNA must be performed while on study treatment and at least every 12 weeks after end of treatment for the entire duration of safety follow-up.
    3. Antiviral prophylaxis must be implemented before the first administration of the study treatment, and continued up to 12 months after end of study treatment. If antiviral therapy cannot be given or if the patient is not willing to comply with the antiviral treatment requirement, the patient is not eligible for the study.
  * Hepatitis C: patients with positive hepatitis C antibody and HCV-RNA at screening are excluded. Chronic hepatitis C patients who have completed HCV anti-viral treatment must be HCV-RNA negative at least 12 weeks after treatment before randomization to be eligible. Cases of spontaneous HCV clearance should be discussed with sponsor before enrollment.
* Evidence of active tuberculosis (TB) infection is exclusionary. Patient with previously treated TB and previously treated or newly diagnosed latent TB may be eligible.
* Pregnant or nursing (lactating) women,
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while on study treatment and for 6 months after stopping of investigational medication.
* Patients with a known history of non-compliance to medication, or who were unable or unwilling to complete PRO questionnaires, or who are unable or unwilling to use the device for collection of PROs.
* United States (and other countries, if locally required): Sexually active males, unless they agree to use barrier protection during intercourse with a woman of childbearing potential, while taking study treatment. As condom use alone has a reported failure rate exceeding 1% per year, it is recommended that female partners of male study participants use a second method of birth control.

Although ianalumab is not teratogenic and/or genotoxic, and not transferred to semen, male contraception is required, as requested by FDA.

Globally, for all sexually active males, contraception should be used in accordance with locally approved prescribing information of concomitant medications administered.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2027-05-13 (Estimated)

PRIMARY OUTCOMES:
Plan A and B - Change from baseline in ESSDAI score at Week 48 | 48 weeks
  * Plan A - United States of America and US reference countries
  * Plan B - EU, China, other non-US Regions and EU reference countries
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status.

SECONDARY OUTCOMES:
Change from baseline in SSSD score at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  The Sjogrens Syndrome Symptom Diary (SSSD) is questionnaire consists of five (six for females) questions about symptoms of Sjögren's syndrome, each question given a score of 0-10 (0=no symptoms, 10=worst possible symptoms) where patient choose the one response that best describes how severe the symptom was at its worst in the PAST 24 HOURS. It includes six symptom items (eye dryness, mouth dryness, skin dryness, physical fatigue, muscle and/or joint pain, genital dryness), and applies a recall period of 24 hrs. The aim of the SSSD is to establish patient reported endpoints for the treatment of Sjogrens syndrome. Participants will complete the diary daily for 7 days prior to the scheduled dosing.
Percentage of participants achieving ESSDAI response at Week 48** | 48 weeks
  Efficacy (Plan A and B)
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status
Percentage of participants achieving ESSDAI score <5 at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  Dose response measured by change multi-dimensional disease activity as assessed by the physician. Score range is 0-123. Higher scores on the EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) scale are associated with poorer health states A negative change from baseline indicates improvement in disease status
Percentage of participants achieving SSSD response at Week 48** | 48 weeks
  Efficacy (Plan A and B)
  The Sjogrens Syndrome Symptom Diary (SSSD) is questionnaire consists of five (six for females) questions about symptoms of Sjögren's syndrome, each question given a score of 0-10 (0=no symptoms, 10=worst possible symptoms) where patient choose the one response that best describes how severe the symptom was at its worst in the PAST 24 HOURS. It includes six symptom items (eye dryness, mouth dryness, skin dryness, physical fatigue, muscle and/or joint pain, genital dryness), and applies a recall period of 24 hrs. The aim of the SSSD is to establish patient reported endpoints for the treatment of Sjogrens syndrome. Participants will complete the diary daily for 7 days prior to the scheduled dosing.
Change from baseline in stimulated whole salivary flow rate at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  Both the amount and composition of saliva has been shown to reflect the glandular damage caused by the disease process of Sjögren's (Pijpe et al 2007). Unstimulated and stimulated salivary secretions are collected over 5 minutes. As much as possible the assessments are to be performed at a fixed time of the day to minimize fluctuations related to the circadian rhythm of salivary flow and composition (Dawes 1972).
Change from baseline in PhGA at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  Physician global assessment of disease activity is made with relation to Sjögren's syndrome. Physician's global assessment (PhGA) of disease activity for Sjögren's syndrome is performed using 3 separate scales:
  * Visual Analog Scale (VAS) - an unnumbered 100 mm long horizontal line ranging from "no disease activity' to "maximal disease activity". The assessment of patient's condition on the day is made by placing a vertical mark across the line.
  * Numerical Rating Scale (NRS) - a segmented numeric version of the VAS. A respondent needs to select a whole number (0-10 integers), with 0 being "no disease activity" and 10 being "maximal disease activity".
  * 4-point Likert scale - The level of disease activity is assessed on a scale from "inactive" to "high activity".
Change from baseline in PaGA at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  Patient's global assessment (PaGA) of disease activity for Sjögren's syndrome is performed using 3 separate scales:
  * Visual Analog Scale (VAS) - an unnumbered 100 mm long horizontal line ranging from "very good' to "very poor". The assessment is made by placing a vertical mark across the line.
  * Numerical Rating Scale - a segmented numeric version of the VAS. A respondent needs to select a whole number (0-10 integers), with 0 being "very poor" and 10 being "very good".
  * 4-point Likert scale - The level of symptom severity is assessed on a scale from "none to severe".
Change from baseline in FACIT-F score at Week 48 | 48 weeks
  Efficacy (Plan A and B)
  The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F version 4) is a short, 13-item, easy-to-administer tool that measures an individual's level of fatigue during their usual daily activities over the past week (Webster et al 2003). The level of fatigue is measured on a 5-point Likert scale (0 = not at all, 1 = a little bit, 2 = somewhat, 3 = quite a bit, 4 = very much).
Change from baseline in ESSPRI score at Week 48 | 48 weeks
  Efficacy (Plan B)
  ESSPRI is an established disease outcome measure for Sjögren's (Seror et al 2011, Seror et al 2015). It consists of three domains of dryness, pain and fatigue.
  The subject assesses severity of symptoms they experience on a single 0-10 numerical scale for each of the three domains. The ESSPRI score is defined as the mean of scores from the three scales: (dryness + pain + fatigue) /3. ESSPRI will be applied to the study patients at during runin period, at baseline and during study treatment.
Percentage of participants achieving ESSPRI response at Week 48** | 48 Weeks
  Efficacy (Plan B)
  ESSPRI is an established disease outcome measure for Sjögren's (Seror et al 2011, Seror et al 2015). It consists of three domains of dryness, pain and fatigue.
  The subject assesses severity of symptoms they experience on a single 0-10 numerical scale for each of the three domains. The ESSPRI score is defined as the mean of scores from the three scales: (dryness + pain + fatigue) /3. ESSPRI will be applied to the study patients at during run-in period, at baseline and during study treatment.

OTHER OUTCOMES:
Incidence of Treatment-emergent AEs (TEAEs) /SAEs (Serious Adverse Event) upto the end of the study | Through study completion up to two years
  Safety(Plan A and B)
Incidence of anti-ianalumab antibodies in serum Anti Drug Antibody (ADA) assay to end of study | through study completion up to 2 years
  Immunogenicity (Plan A and B)
Ianalumab concentration in serum during the treatment and follow-up (up to the end of study) | throughout study completion up to 2 years
  Pharmacokinetics (Plan A and B)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (134):
- United States (23):
  - Providence Medical Foundation, Fullerton, California
  - Advanced Medical Research, La Palma, California
  - Bay Area Arthritis And Osteoporosis, Brandon, Florida
  - GNP Research, Cooper City, Florida
  - Sarasota Arthritis Res Ctr, Sarasota, Florida
  - Augusta University Georgia, Augusta, Georgia
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - Clin Invest Specialists Inc, Orland Park, Illinois
  - Clinic of Robert Hozman, Skokie, Illinois
  - Clinical Investigation Specialists, Inc., Wauconda, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Tufts School of Dental Medicine, Boston, Massachusetts
  - Arthritis Osteoporosis Assoc of NM, Las Cruces, New Mexico
  - St Lawrence Health System, Potsdam, New York
  - On Site Clinical Solutions Llc, Charlotte, North Carolina
  - Arthritis and Osteoporosis, Charlotte, North Carolina
  - RAO Research LLC, Oklahoma City, Oklahoma
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C Gupta MD Memphis TN, Memphis, Tennessee
  - Prolato Clinical Research Center, Houston, Texas
  - First Outpatient Research Unit, San Antonio, Texas
  - Advanced Rheumatology of Houston, Spring, Texas
  - Arthritis Northwest PLLC, Spokane, Washington
- Argentina (4):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Miguel Tucuman, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
- Australia (3):
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Woodville South, South Australia
  - Novartis Investigative Site, Hobart, Tasmania
- Brazil (3):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (3):
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (6):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Sydney, Nova Scotia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Rimouski, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Chile (3):
  - Novartis Investigative Site, Concepción, Bio Bio
  - Novartis Investigative Site, Valdivia, Los Ríos Region
  - Novartis Investigative Site, Santiago, RM
- China (15):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Yinchuan, The Ningxia Hui Autonomous Reg
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Xinxiang
- Colombia (4):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
- France (5):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Strasbourg
- Germany (5):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Herne
- Novartis Investigative Site, Athens, Greece
- Hungary (5):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Szeged
- India (4):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi
- Israel (2):
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
- Italy (5):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Napoli
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kuwana, Mie-ken
  - Novartis Investigative Site, Sasebo, Nagasaki
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Meguro-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
- Mexico (3):
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Mérida, Yucatán
  - Novartis Investigative Site, México
- Poland (5):
  - Novartis Investigative Site, Poznan, Greater Poland Voivodeship
  - Novartis Investigative Site, Krakow, Lesser Poland Voivodeship
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Romania (3):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
- Slovakia (4):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Partizánske
  - Novartis Investigative Site, Zvolen
- South Africa (2):
  - Novartis Investigative Site, Panorama, Western Cape
  - Novartis Investigative Site, Stellenbosch, Western Cape
- Spain (6):
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Stockholm, SE, Sweden
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
- United Kingdom (5):
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Swindon

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com